CLINICAL TRIAL: NCT03219684
Title: A Descriptive Study on the Effectiveness and Safety of Cyclosporin A Therapy in Steroid Dependent and Steroid Resistant Childhood Nephrotic Syndrome
Brief Title: Cyclosporin A Therapy in Childhood Nephrotic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdullah Ahmed Abdel_Ghany, principal investigator, Assiut University
Other Study IDs: DSESCSDSRNS
Record Dates: First submitted 2017-07-11; First posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Steroid Dependent and Steroid Resistent Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Diagnostic Test: serum protein ,kidney function ,liver function.,serum cholesterol — monthly review of serum protein kidney function ,liver function and serum cholesterol in all patients

SUMMARY:
Nephrotic syndrome (NS) is among the most common pediatric kidney diseases and is defined as massive proteinuria (>40 mg/m2/h or urine protein to creatinine ratio >2 g/g) leading to hypoalbuminemia (<2.5 g/dL), edema, and hyperlipidemia. 60-70 % of patients present prior to age of 6 years

DETAILED DESCRIPTION:
. Most children with NS are treated initially with oral corticosteroids, and they can be clinically classified based on their ability to achieve remission (i.e., complete normalization of proteinuria). Approximately 85 % of children under the age of 6 years are steroid-sensitive, whereas the remainder have steroid-resistant disease. Older children are more likely to have steroid-resistant NS. Children with steroid-resistant disease may have an underlying genetic cause for NS, and providers should consider genetic testing in this population, depending on the age of the child . While inherited causes of NS are often resistant to all therapies, there are reports of complete or partial remission in some children .

For those children who respond to steroids, the majority will have one or more relapses and half will have frequently relapsing (≥4 relapses/year) or steroid-dependent (two consecutive relapses during steroid therapy or within 14 days of stopping steroids). NS Children with frequently relapsing NS and steroid-dependent NS may have significant side effects from cumulative corticosteroid therapy so treatment with other agents is often required .

Cyclosporine and tacrolimus are calcineurin inhibitors that are commonly used as immunosuppressive agents in solid organ transplantation. CNIs are recommended as first-line therapy for children with steroid-resistant NS and as steroid-sparing agents for children with frequently relapsing or steroid-dependent NS .Calcineurin inhibitors (CNIs) inhibit T-cell activation and may be exerting their effect in nephrotic syndrome through this mechanism.

Alternately, cyclosporine has been shown to directly target the podocyte and stabilize the actin cytoskeleton responsible for maintaining cell shape(5) .. Although the majority of studies in nephrotic syndrome have been performed with cyclosporine, tacrolimus appears to be equally efficacious.

Cyclosporin A therapy is well recognised regarding its steroid sparing effect in steroid dependant patients and is responsible for maintaining remission in more than 75% of patients with Steroid dependent nephrotic syndrome even after discontinuation of steroids Furthermore, it has been shown to be effective in inducing remission in steroid resistant nephrotic syndrome. However ,Cyclosporin A is associated with a plethora of side effects such as hypertension, nephrotoxicity hypertrichosis, gum hyperplasia, gastrointestinal disturbances and tremor.

ELIGIBILITY:
Inclusion Criteria:

* The study will include all children (on cyclosporine therapy for treatment of Steroid dependent or Steroid resistant nephrotic syndrome ) who present to Nephrology Unit , and clinic at Assiut University Children Hospital during one year duration.

Exclusion Criteria:

* children with adequate response to steroid therapy and without relapses or resistance to steroid therapy

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children from the age of one year to the age of 18 year who are diagnosed as steroid resistent and steroid dependent nephrotic syndrome and on cyclosporin therapy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of nephrotic state of each patient for evaluation of efficacy of cyclosporin A therapy | one year
  measurment of serum albumin ,serum cholesterol and urinary protien excretion
evaluation of side effects of cyclosporin A | one year
  serial observation of common side effects of cyclosporin A as hypertension, nephrotoxicity hypertrichosis, gum hyperplasia, gastrointestinal disturbances and tremor.

IPD SHARING:
Plan to Share IPD: Undecided